CLINICAL TRIAL: NCT02727491
Title: A Prospective Randomized Double-blind Placebo Controlled Trial; Does Pre and Postoperative Dextromethorphan Reduce Post-tonsillectomy Pain in Children?
Brief Title: Does Pre and Postoperative Dextromethorphan Reduce Post-tonsillectomy Pain in Children?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Rachel Rooney (Other)
Responsible Party: Sponsor-Investigator, Dr. Rachel Rooney, Dr. Rachel Rooney, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANAE-182-10
Record Dates: First submitted 2016-02-11; First posted 2016-04-04 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Pain, Postoperative
Keywords: opioid analgesics,; opioid consumption; adverse effects; postoperative pain; tonsillectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dextromethorphan (Experimental): 1 mg/kg of dextromethorphan syrup orally 30 min preoperatively and then again 8 hours post-tonsillectomy
  Interventions: Drug: Dextromethorphan
- Placebo (Placebo Comparator): 30 min preoperatively and then again 8 hours postoperatively, received inactive placebo syrup identical in volume, appearance and taste as the experimental group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dextromethorphan — Dextromethorphan is a drug of the morphinan class with sedative, dissociative, and stimulant properties (at higher doses). Dextromethorphan has been explored for a number other uses in medicine, including pain relief (as either the primary analgesic, or an opioid potentiator).
  Other Names: dextromethorphan hydrobromide
  Arms: dextromethorphan
Drug: Placebo — Placebo syrup identical to active comparator in taste, appearance and volume but is inactive. Placebo comparator will be used in the placebo arm of the trial.
  Other Names: control
  Arms: Placebo

SUMMARY:
With Institutional ethics board and Health Canada approval, pediatric patients (ages 3-12) undergoing tonsillectomy or adenotonsillectomy (under standardized anesthesia) will be randomized to receive dextromethorphan hydrobromide (1mg/kg orally) 30 min preoperatively and again 8 hours postoperatively OR placebo (syrup identical in taste, appearance and volume) at the same time points. The primary outcome is an integrated assessment of perioperative pain scores and opioid use for 24 hours postoperatively. Secondary outcomes include nausea, vomiting, respiratory depression, and bleeding for 24 hours postoperatively. Our hypothesis is that dextromethorphan will decrease the incidence/severity of post-tonsillectomy pain. The improved pain control will be apparent through reduced opioid consumption and integrated pain scores. This will result in a reduced incidence of opioid-related side effects and adverse events.

DETAILED DESCRIPTION:
With Institutional ethics board and Health Canada approval and parental consent and child assent, pediatric patients (ages 3-12) undergoing tonsillectomy or adenotonsillectomy (under standardized anesthesia) will be randomized to receive dextromethorphan hydrobromide (1mg/kg orally) 30 min preoperatively and again 8 hours postoperatively OR placebo (syrup identical in taste, appearance and volume) at the same time points. The primary outcome is an integrated assessment of perioperative pain scores and opioid use for 24 hours postoperatively. Pain scores were collected preoperatively at rest and then at 1,2,3,8,9,10 and 24 hours postoperatively using the validated Children's Hospital of Eastern Ontario Pain Scale (CHEOPS). Secondary outcomes include nausea, vomiting, respiratory depression, and bleeding recorded by blinded observers for 24 hours postoperatively.

Our hypothesis is that dextromethorphan will decrease the incidence/severity of post-tonsillectomy pain. The improved pain control will be apparent through reduced opioid consumption and integrated pain scores. This will result in a reduced incidence of opioid-related side effects and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's (ASA) physical classification I and II
* tonsillectomy or adenotonsillectomy
* admission to extended postoperative care unit

Exclusion Criteria:

* use of monoamine oxidase inhibitors, serotonin reuptake inhibitors or tricyclic antidepressants
* requirement of preoperative sedation
* recent dextromethorphan use (<24 h before surgery)
* intolerance, sensitivity or contraindication to any agents used in the study
* pre-existing chronic pain or chronic analgesic use
* body mass index (BMI) for age percentile greater than 90
* confounding procedural factors which might affect the validity of the data
* inability to adhere to study protocol
* contraindication to volatile anesthetics

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
integrated assessment of pain scores and opioid use | 24 hours postoperatively
  The Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) will be measured at rest 24 hours postoperatively and this will be integrated with total opioid consumption at 24 hours postoperatively. This will be achieved by converting both pain scores and opioid consumption to % change. The % differences for each of the 2 variables are then added together on a per-subject basis to provide a summated % difference. The individual and summated % differences can then be plotted on a single graph and the integrated ranks of the experimental and control groups can be compared with standard statistical tests.(1)

SECONDARY OUTCOMES:
opioid-related adverse effects | up to 24 hours postoperatively
  nausea, vomiting, respiratory depression, bleeding
pain scores | 1,2,3,8,9 and 10 hours postoperatively
  Pain scores at rest on the CHEOPS pain scale

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Rooney, MD, FRCPC, Principal Investigator — Queen's University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silverman DG, O'Connor TZ, Brull SJ. Integrated assessment of pain scores and rescue morphine use during studies of analgesic efficacy. Anesth Analg. 1993 Jul;77(1):168-70. No abstract available. PMID 8317727
- [Background] Kawamata T, Omote K, Kawamata M, Namiki A. Premedication with oral dextromethorphan reduces postoperative pain after tonsillectomy. Anesth Analg. 1998 Mar;86(3):594-7. doi: 10.1097/00000539-199803000-00031. PMID 9495423
- [Background] Dawson GS, Seidman P, Ramadan HH. Improved postoperative pain control in pediatric adenotonsillectomy with dextromethorphan. Laryngoscope. 2001 Jul;111(7):1223-6. doi: 10.1097/00005537-200107000-00015. PMID 11568544
- [Background] Kelly LE, Sommer DD, Ramakrishna J, Hoffbauer S, Arbab-Tafti S, Reid D, Maclean J, Koren G. Morphine or Ibuprofen for post-tonsillectomy analgesia: a randomized trial. Pediatrics. 2015 Feb;135(2):307-13. doi: 10.1542/peds.2014-1906. PMID 25624387
- [Background] Hasan RA, Kartush JM, Thomas JD, Sigler DL. Oral dextromethorphan reduces perioperative analgesic administration in children undergoing tympanomastoid surgery. Otolaryngol Head Neck Surg. 2004 Nov;131(5):711-6. doi: 10.1016/j.otohns.2004.06.709. PMID 15523452
- [Background] Rose JB, Cuy R, Cohen DE, Schreiner MS. Preoperative oral dextromethorphan does not reduce pain or analgesic consumption in children after adenotonsillectomy. Anesth Analg. 1999 Apr;88(4):749-53. doi: 10.1097/00000539-199904000-00012. PMID 10195517
- [Background] Weinbroum AA, Rudick V, Paret G, Ben-Abraham R. The role of dextromethorphan in pain control. Can J Anaesth. 2000 Jun;47(6):585-96. doi: 10.1007/BF03018952. PMID 10875724
- [Background] Brown KA, Laferriere A, Lakheeram I, Moss IR. Recurrent hypoxemia in children is associated with increased analgesic sensitivity to opiates. Anesthesiology. 2006 Oct;105(4):665-9. doi: 10.1097/00000542-200610000-00009. PMID 17006062
- [Background] Steinberg GK, Bell TE, Yenari MA. Dose escalation safety and tolerance study of the N-methyl-D-aspartate antagonist dextromethorphan in neurosurgery patients. J Neurosurg. 1996 May;84(5):860-6. doi: 10.3171/jns.1996.84.5.0860. PMID 8622162